CLINICAL TRIAL: NCT03428841
Title: Audiovisual Assessment After Dural Puncture During Epidural Placement in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 18-02
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Hearing Loss
Keywords: audiometry; dural puncture; epidural
MeSH Terms: conditions — Hearing Loss | interventions — Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with dural puncture at epidural: Patients who sustained an accidental dural puncture during the epidural procedure.
  Interventions: Procedure: Audiometry
- Patients with no dural puncture: Patients with no dural puncture during epidural procedure, to serve as a control group.
  Interventions: Procedure: Audiometry

INTERVENTIONS:
Procedure: Audiometry
  Other Names: hearing test

SUMMARY:
The study involves assessment of hearing and visual complications along with headache after accidental dural puncture in patients receiving epidurals. Hearing loss will be assessed by clinical examination and audiometry testing, while visual complications will be assessed by clinical examination. The patients will receive standard treatment for headache in the form of drugs and if required an epidural blood patch ( injecting patient's blood in the epidural space). The course of these complications and response to treatment will be investigated over a period of time.

Audiometry results from patients with dural puncture will be compared to those of patients who also had epidurals, but without a dural puncture.

The investigators hypothesize that audiovisual complications occur more frequently in patients having accidental dural puncture with epidural needle and that the symptoms resolve with the administration of epidural blood patch.

DETAILED DESCRIPTION:
Although many studies have reported auditory complications after spinal, none have been done in obstetric patients with accidental dural puncture with epidural needle. Long term follow up of these complications has been unknown. The incidence of both auditory and visual complications is likely to be high in patients getting accidental dural puncture with 17G Touhy epidural needle as compared to small gauge spinal needles. Several case reports have been reported with such temporary and permanent hearing and visual loss. A prospective study to understand these complications is required. The study will provide us with the true incidence of audiovisual complications of dural puncture with an epidural needle. Early intervention in cases of dural puncture may alleviate or halt symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Parturients having accidental dural puncture during epidural placement for labour analgesia.
* Patients who give written informed consent to participate in the study.
* Dural puncture with 17G Touhy needle with/out headache
* Postural headache after 24 hours of epidural
* Labouring women undergoing vaginal or Cesarean delivery
* For the control group, patients with no dural puncture during epidural placement

Exclusion criteria:

* Patients refusing to consent
* Dural puncture with spinal needle

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women having epidural analgesia for labour pain management.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-09-25 (Actual); Primary Completion 2010-02-18 (Actual); Study Completion 2010-04-30 (Actual)

PRIMARY OUTCOMES:
Hearing loss | 1 month
  Hearing loss as measured by audiometry

SECONDARY OUTCOMES:
Severity of headache | 1 month
  Pain from postdural puncture headache, rated on verbal numeric rating scale (VNRS) from 0-10, where 0 represents no pain and 10 represents worst pain.
Associated vestibular symptoms | 1 month
  The presence of nausea, vomiting, vertigo, dizziness, associated with the dural puncture headache.
Associated cochlear symptoms | 1 month
  The presence of hearing loss, hyperacusis or tinnitus, associated with the dural puncture headache.
Ocular symptoms | 1 month
  The presence of photophobia, teichopsia, diplopia or difficulty in accommodation, associated with the dural puncture headache.
Musculoskeletal symptoms | 1 month
  The presence of neck stiffness or scapular pain, associated with the dural puncture headache.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada